CLINICAL TRIAL: NCT03728465
Title: An Open Label Phase II Study to Evaluate Safety and Efficacy of Combined Treatment With Ipilimumab and Nivolumab in Patients With Four and More Symptomatic Brain Metastases of Melanoma
Brief Title: Evaluation of Safety and Efficacy of Patients With Four and More Symptomatic Brain Metastases of Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-429
Record Dates: First submitted 2018-10-19; First posted 2018-11-02 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Melanoma; Brain Metastases
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Phase (Experimental): Treatment phase is divided into the "Induction Phase" and "Maintenance Phase". During the induction phase patients are treated with 1 mg/kg nivolumab and 3 mg/kg ipilimumab, during the maintenance phase with nivolumab 3 mg/kg only .
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — In the induction phase of this study nivolumab is administered as a IV infusion in combination with ipilimumab at a dose of 1 mg/kg for 4 cycles at three weeks interval and in a maintenance phase alone at a dose of 3 mg/kg every two weeks.
  Other Names: OPDIVO
Biological: Ipilimumab — In the induction phase of this study ipilimumab is administered as a IV infusion in combination with nivolumab at a dose of 3 mg/kg for 4 cycles at three weeks interval.
  Other Names: YERVOY

SUMMARY:
Up to 50% of patients with unresectable metastatic melanoma will develop brain metastases during their lifetime. A possible treatment options for patients with brain metastases are surgery and radiotherapy but usually for lesions in the range of < 3 brain metastases. This study was performed to evaluate the addition of immune checkpoint inhibitors in patients with stage IV melanoma with > 3 symptomatic brain metastases, who are not eligible for surgery or radiosurgery.

DETAILED DESCRIPTION:
Brain metastases are a frequent problem in patients with melanoma. Up to 50% of patients with unresectable metastatic melanoma will develop brain metastases during their lifetime with a median overall survival of 4 months. Surgical removal or stereotactic radiosurgery of brain metastases can improve overall survival in patients with a limited number of lesions, usually in the range of one to three brain metastases depending on neuroanatomical localization. This benefit is no longer present when considering patients with > 3 brain metastases. As cytotoxic chemotherapy and multiple chemotherapeutic agents show only limited activity in > 3 brain metastases patients, immune checkpoint inhibitors such as ipilimumab and nivolumab offer new opportunities to improve disease outcomes for these patients.

This open label phase II study evaluates safety and efficacy of combined treatment with ipilimumab and nivolumab in patients with stage IV melanoma with four or more symptomatic brain metastases, who are not eligible for surgery or radiosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (ICF) prior to any screening procedures being performed
* Ability to comply with protocol requirements
* Metastatic histologically confirmed melanoma that is unresectable
* Presence of > 3 active brain metastases confirmed/evaluated by MRI
* Measurable disease by MRI per iRANO and RECIST 1.1 criteria
* The time between the baseline MRI and the date of registration should not exceed 28 days. Steroid treatment is permissible before brain MRI evaluation but the dose should have been stable for at least 7 days and should be carefully documented
* Patient must agree to the cerebro-spinal fluid (CSF) collections according to the study protocol
* Patients naïve for systemic treatment are eligible
* Patients pretreated with systemic immunotherapy, targeted therapy or chemotherapy are eligible (exception: previous treatment with the combination of CTLA-4 and PD-1 antibodies)
* Patients must have recovered completely from any treatment-related acute toxicity associated with prior therapy
* At least two weeks must have passed since the last systemic anti-cancer treatment
* Patients with prior local therapy of brain metastases are eligible
* Patients may have received irradiation therapies: A) None; B) Whole brain irradiation only, C) Stereotactic irradiation of single or few metastases, D) Combined B+C)
* Screening laboratory values within 14 days prior to registration must meet the criteria: WBC ≥ 2,000/μL, Neutrophils ≥ 1,500/μL, Platelets ≥ 100 x103/μL, Hemoglobin > 9.0 g/dL, Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min, AST/ALT ≤ 3 x ULN, total bilirubin ≤ 1.5 x ULN (except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL), INR ≤ 1.5
* ECOG Performance Status 0, 1 or 2
* Expected life expectancy of ≥ 3 months
* Males and females ≥ 18 years old
* Negative serum pregnancy test within 24 hours prior to the start of study drug for women of childbearing potential (WOCBP)
* Women must not be breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception, as indicated in the ICF, throughout the study and for 23 weeks after the last dose of investigational drug
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception, as indicated in the ICF, throughout the study and for a period of 31 weeks after the last dose of investigational drug. In addition, male patients must be willing to refrain from sperm donation during this time
* Azoospermic males are exempt from contraceptive requirements. WOCBP who are permanently not heterosexually active are also exempt from contraceptive requirements, but must still undergo pregnancy testing as previously described.
* Patients must agree to use at least two methods of contraception, with at least one highly effective method as listed in the ICF

Exclusion Criteria:

* Diagnosed ocular melanoma
* Previous systemic therapy with the combination of CTLA-4 and PD-1 antibodies
* Use of any investigational or non-registered product within the 30 days before registration in the study
* Prior active malignancy within the previous 3 years except locally curable cancers that have been apparently cured, such as: basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix, or breast
* History of organ transplantation
* Active infection requiring systemic therapy
* Active, known or suspected autoimmune disease (exceptions: patients with controlled Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders not requiring systemic treatment).
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Any serious or uncontrolled medical disorders thatmay increase the risk associated with study participation or study drug administration, impair the ability of the patient to receive protocol therapy, or interfere with the interpretation of study results in the opinion of the investigator
* Known substance abuse or psychiatric disorders that would preclude cooperation with tany requirements of the trial
* Legal incapacity or limited legal capacity
* Administration of live, attenuated vaccine within 4 weeks prior to the start of study drug
* Positive test for HBs Ag or HCV antibody
* Known history of a positive test for HIV or known AIDS
* Patients with known allergy or hypersensitivity to any of the study drugs or excipients
* Patients with results of imaging or radiological examinations indicating increased cerebral pressure which would prevent lumbar puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Intracranial Control Rate after 6 months of treatment | 6 months
  Proportion of patients with complete intracranial responses (CR), partial intracranial responses (PR) or stable intracranial disease (SD) after 6 months of treatment.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Number of patients who stay alive after 2 years.
Progression-free survival | 2 years
  Number of patients without progression after 2 years.
Stereotactic irradiation or surgery of brain metastases after partial tumor remission | 2 years
  Percentage of patients in whom stereotactic irradiation or surgery of all metastases becomes applicable after partial tumor remission.
Tolerability according to NCI-CTCAE-Criteria | 2 years
  All adverse events of all grades.
Best Overall Response Rate with Complete Respone (CR) | 6 months
  Percentage of patients with CR at six months of treatment.
Best Overall Response Rate with Partial Response (PR) | 6 months
  Percentage of patients with PR at six months of treatment.
Cognitive function evaluation by standardized diagnostic procedures | 2 years
  Systemic longitudinal neuropsychological evaluation to investigate the influence of therapy on cognitive performance will be performed by standardized diagnostic procedures.
Quality of life evaluation with RAND 36-Item Health Survey 1.0 | 2 years
  Quality of life assessment is evaluated with the RAND 36-Item Health Survey questionnaires which include physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Evaluation will be performed according to the manual.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, Prof.Dr.med., Principal Investigator — University Hospital Tuebingen
Locations (11):
- Germany (11):
  - Elbe Kliniken Stade - Buxtehude GmbH, Buxtehude
  - Universitätsklinik Carl Gustav Carus Dresden, Dresden
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Gesellschaft für Klinische Forschung Ludwigshafen mbH, Ludwigshafen
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum rechts der Isar, München
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No